CLINICAL TRIAL: NCT06634394
Title: A Phase 1b/2 Open-Label Study of APVO436 in Combination With Venetoclax and Azacitidine in Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: APVO436 Phase 1b/2 Study in Patients With Newly Diagnosed AML
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aptevo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APVO436-5201
Record Dates: First submitted 2024-10-04; First posted 2024-10-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Arm APVO436 in combination with Venetoclax and Azacitidine (Experimental): APVO436 at escalating dose levels in combination with venetoclax and azacitidine (ven/aza) in adult patients with newly diagnosed, CD123+ AML.
  Interventions: Drug: APVO436; Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: APVO436 — Infusion drug administered as a 4 hour infusion.
Drug: Venetoclax — Oral tablet given on days 1 through 22, of a 28 day cycle.
  Other Names: venclexta
Drug: Azacitidine — Intravenous infusion given on days 1-8 of a 28 day cycle
  Other Names: vidaza

SUMMARY:
A multi-center, open-label, dose-finding study of five dose levels of APVO436 in combination with venetoclax and azacitidine (ven/aza) in adult patients with newly diagnosed, CD123+ AML.

DETAILED DESCRIPTION:
Phase 1b consists of 28-day cycles of treatment in five sequential cohorts. In Cycle 1 (C1) only, to reduce the risk of CRS, each cohort will receive 4 priming doses of APVO436 respectively. APVO436 will be given in combination with venetoclax and azacitidine. For C1D15 and all doses in each subsequent cycle, cohorts will receive APVO436 at the determined cohort dose level.

APVO436 dosing will be administered by a 4-hour intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years. 2. Patient must have confirmation of AML based on 2016 World Health Organization (WHO) criteria and not been previously treated.

  3. Patients must have CD123-positive AML as confirmed by local flow cytometry (or immunohistochemistry [IHC]). Confirmation at diagnosis is acceptable.

  4. Patient must be considered ineligible for induction therapy defined by at least one of the following:
  1. ≥75 years of age
  2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 2 or 3
  3. Cardiac disorder (e.g., congestive heart failure requiring treatment, ejection fraction ≤ 50%, or chronic stable angina)
  4. Pulmonary disorder (e.g., DLCO ≤65% or FEV1 ≤65%)
  5. Creatinine clearance 30-45 mL/min based on Cockcroft-Gault or Modified of Diet in Renal Disease (MDRD) formular
  6. Hepatic disorder with total bilirubin between 1.5 and 3 times the ULN 5. Patient must have a projected life expectancy of ≥12 weeks

Exclusion Criteria:

1. Patient has received treatment with the following:

   1. A hypomethylating agent, venetoclax, and/or chemotherapeutic agent for AML, myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), or myelodysplastic/myeloproliferative neoplasms (MPS/MPN)
   2. CAR-T cell therapy or history of allogeneic hematopoietic stem cell transplant (HSCT)
   3. Experimental therapies for MDS or AML
2. Patient is currently participating in another interventional research study.
3. Patient has history of MPN including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia (CML) with or without BCR-ABL1 translocation, or AML with BCR-ABL1 translocation.
4. Patient has acute promyelocytic leukemia.
5. Patient has a current autoimmune disorder requiring immunosuppressive therapy such as systemic (oral or IV) steroid therapy >10 mg methylprednisolone daily or its equivalent
6. Patient is receiving concurrent corticosteroid therapy as an anticancer drug (any dose).
7. Patient has known active CNS involvement with AML. Patients who received intrathecal chemotherapy for prophylaxis of AML in the CNS prior to enrollment may enroll in this study.
8. Creatinine clearance <30ml/min based on Cockcroft-Gault or MDRD formular.
9. Bilirubin of >3xULN in the absence of Gilbert's Syndrome.
10. AST and/or ALT >3 times the ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
To assess the safety, tolerability, and maximum tolerated dose (MTD) of increasing doses of APVO436 in combination with venetoclax/azacitidine in patients with newly diagnosed AML | Through the end study completion average of 1 year.
  Incidence and severity of treatment emergent adverse events (TEAEs), including ≥Grade 3 adverse events (AEs), serious AEs (SAEs), and AEs of special interest (AESIs: ≥Grade 2 infusion related reaction (IRR), ≥Grade 2 cardiac toxicity, and ≥Grade 2 neurotoxicity as complication of cytokine release syndrome [CRS]).

SECONDARY OUTCOMES:
Determine the efficacy of increasing doses of APVO436 in combination with venetoclax and azacitidine in patients with newly diagnosed AML | Through the end study completion average of 1 year.
  Complete remission (CR) rate

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Huebner, MD, Study Director — Aptevo Therapeutics
Locations (7):
- United States (7):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami, Miami, Florida
  - University of Kansas, Fairway, Kansas
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided